CLINICAL TRIAL: NCT04458688
Title: Investigating the Effect of Ocrelizumab in African Americans and Caucasians With Relapsing Multiple Sclerosis: a Novel, Advanced Multimodal MRI and Optical Coherence Tomography-Angiography (OCTA) Study
Brief Title: Investigating the Effect of Ocrelizumab in African Americans and Caucasians With Relapsing Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Evanthia Bernitsas, MD, Prinipal Investigator, Wayne State University
Other Study IDs: ML41569
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: multiple sclerosis; ocrelizumab; magnetic resonance imaging (MRI); optical coherence tomography angiography (OCTA)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- African Americans with RRMS: Participants who are diagnosed with relapsing multiple sclerosis and who have chosen to start or recently started using ocrelizumab as their disease modifying therapy. Age range: 18 to 60 years old. Ethnicity: Self-described as African American.
  Interventions: Other: Observation of Ocrelizumab as Treatment in RRMS Patients
- Caucasian American with RRMS: Participants who are diagnosed with relapsing multiple sclerosis and who have chosen to start or recently started using ocrelizumab as their disease modifying therapy. Age range: 18 to 60 years old. Ethnicity: Self-described as Caucasian American.
  Interventions: Other: Observation of Ocrelizumab as Treatment in RRMS Patients

INTERVENTIONS:
Other: Observation of Ocrelizumab as Treatment in RRMS Patients — It is decided by the patient and their physician to begin taking ocrelizumab PRIOR to study enrollment. The study is only observing the effects of ocrelizumab as a pre-decided treatment option for a patient's MS.
  Other Names: Observing Ocrelizumab Use

SUMMARY:
The investigators intend to examine the effects of ocrelizumab use in African American multiple sclerosis disease course compared to Caucasian disease course utilizing imaging measures with magnetic resonance imaging (MRI) and optical coherence tomography angiography (OCT-A)..

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a disease of the central nervous system (CNS). Several lines of evidence suggest that MS is an autoimmune disease with both T and B-cell activity leading to CNS inflammation which results in demyelinating injury. Ocrelizumab was FDA approved in March 2017 for relapsing remitting (RRMS) and primary progressive multiple sclerosis (PPMS) by depleting B cells. It has shown to be effective in reducing the annualized relapse rate, decreasing disability progression, and reducing the number of new and active MRI brain lesions.

Previous research studies have reported a more aggressive course in African Americans with MS, more lesions on the MRI scan, and more severe injury to layers of the eye (specifically in the retina) compared to Caucasians.

This is a novel study investigating the effect of ocrelizumab in African American relapsing multiple sclerosis (RMS) patients compared to Caucasian RMS patients using imaging measures, specifically multimodal magnetic resonance imaging (MRI) and optical coherence tomography-angiography (OCTA). This is a non-drug intervention study; therefore, patients who are recruited will have already decided to make ocrelizumab their disease-modifying therapy before enrollment. The study will recruit 86 (including 6 potential screen fails) patients in total (40 African American patients and 40 Caucasian patients who are matched by age, sex, disease duration, and disease disability. The study will consist of 5 visits in six-month intervals across two years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have chosen to start ocrelizumab and for whom ocrelizumab is determined to be the most appropriate standard-of-care disease modifying therapy (DMT) by the treating neurologist.
2. May be treatment naive, or had suboptimal response to no more than one DMT after an adequate course of treatment (defined as treatment duration of 6+ months).
3. Age 18 to 60 years old.
4. Ethnicity: self-identified as African American or Caucasian.
5. Clinically definite relapsing remitting multiple sclerosis (RRMS) per 2017 revised McDonald criteria.
6. EDSS from 0 to 6 (inclusive) at baseline visit.
7. Able to give informed consent.
8. Able to have MRI scans.

Exclusion Criteria:

1. Treatment with another monoclonal antibody, including but not limited to natalizumab, alemtuzumab, daclizumab.
2. Failed 2 or more DMTs.
3. Treatment with immunosuppressant agents, such as chemotherapeutic agents.
4. Claustrophobia.
5. Allergy to contrast.
6. Significant medical problems that the PI determines will interfere with the conduct of the study.
7. Relapse or use of corticosteroids within 30 days prior to baseline visit.
8. Pregnancy.
9. History of kidney or liver insufficiency.
10. History of malignancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants who are diagnosed with relapsing multiple sclerosis and who have chosen to start or recently started using ocrelizumab as their disease modifying therapy. Age range: 18 to 60 years old. Ethnicity: self-described as African American or Caucasian.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) with contrast | Change in MRI at BL, Month 6, Month 12, and Month 24
  Approximately a 1 hour MRI with contrast (administered via IV)
Optical Coherence Tomography Angiography (OCTA) | Change in OCTA at BL, Month 12, and Month 24
  Eye scan with contrast (administered via IV)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Bernitsas, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, ICFs, study reports, statistical analysis plans, secure CRFs, and results will be shared with Roche/Genentech Inc. All patient data will have a unique number/digit code when sent to protect patient identity.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for the duration of the study and up to 15 years after the last patient has completed the study.
Access Criteria: All data will be stored and shared in electronic case report form (eCRF) format.